CLINICAL TRIAL: NCT03127969
Title: Is Fluidotherapy Effective in Rheumatoid Hand? A Randomized Controlled Trial
Brief Title: Is Fluidotherapy Effective in Rheumatoid Hand?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selmin Gulbahar (Other)
Responsible Party: Sponsor-Investigator, Selmin Gulbahar, Clinical Professor and Head of Department of Physical Medicine and Rehabilitation, Faculty of Medicine, Dokuz Eylul University, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DorkuzEUftr1
Record Dates: First submitted 2017-04-04; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid hand; Fluidotherapy; Rehabilitation
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Fluidotherapy treatment (Other): Patients who received fluidotherapy and joint protection and exercise
  Interventions: Other: Fluidotherapy treatment; Other: Joint protection and exercise
- Joint protection and exercise (Other): Patients who received joint protection and exercise
  Interventions: Other: Joint protection and exercise

INTERVENTIONS:
Other: Fluidotherapy treatment — fluidotherapy and joint protection and exercise
  Arms: Fluidotherapy treatment
Other: Joint protection and exercise — joint protection and exercise

SUMMARY:
The objective of this study is to evaluate the efficacy of fluidotherapy primarily on function and quality of life, secondarily on pain, morning stiffness, grip strength, and disease activity in patients with rheumatoid hand.Ninety-three patients were enrolled in this prospective, single-blind, randomized, and controlled trial. Patients were randomized into 2 groups. Group 1 (n=47) had fluidotherapy (5 times per week, for 3-week duration) and Group 2 (n=46) was the control group. All patients received joint protection and exercise program. The primary outcome measures were Health Assessment Questionnaire (HAQ) and Duruöz Hand Index (DHI) and secondary outcome measures were pain and morning stiffness assessed using the Visual Analog Scale (VAS, 0-100 mm), the Grip Ability Test (GAT), Disease Activity Score-28 (DAS-28), and grip strength. These assessments were performed at baseline, at week 3 and week 12 after treatment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-75 years RA diagnosis fulfilling ACR 2010 criteria
* disease duration for at least 6 months
* no high disease activity and no acute arthritis in the hand according to DAS-28
* hand problem specified with pain and loss of function in the hand
* being in an eligible sociocultural and socioeconomic state so as to be able to come to the ambulatory treatment program

Exclusion Criteria:

* change of medication within the last 3 months or during the study (except for non-steroidal anti-inflammatory drugs and paracetamol)
* changes in oral corticosteroid dose in the last month, intraarticular or intramuscular corticosteroid use
* hand or upper extremity surgery in the last 6 months
* previous injury in the hand or upper extremity in the last 6 months
* pregnancy
* presence of sensory defects in the hand
* presence of cognitive and/or psychiatric disease
* physical therapy for the hand in the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2013-06-18 (Actual); Study Completion 2013-06-18 (Actual)

PRIMARY OUTCOMES:
Health Assessment Questionnaire (HAQ) | Change from Baseline, Health Assessment Questionnaire score at 3 weeks and 12 weeks
Duruöz Hand Index (DHI) | Change from Baseline. Duruöz Hand Index score at 3 weeks and 12 weeks

SECONDARY OUTCOMES:
pain | baseline, at week 3 and week 12
  Visual Analog Scale (VAS, 0-100 mm)
stiffness | baseline, at week 3 and week 12
  Visual Analog Scale (VAS, 0-100 mm)
Grip Ability Test (GAT) | baseline, at week 3 and week 12
Disease Activity Score-28 (DAS-28) | baseline, at week 3 and week 12
grip strength | baseline, at week 3 and week 12
  Jamar measure

IPD SHARING:
Plan to Share IPD: No